CLINICAL TRIAL: NCT00057980
Title: Phase I/II Study of Epirubicin and Celecoxib for Hepatocellular Carcinoma
Brief Title: Epirubicin and Celecoxib in Treating Patients With Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NU 02I6; NU-02I6
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Liver Cancer
Keywords: advanced adult primary liver cancer; localized unresectable adult primary liver cancer; adult primary hepatocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Celecoxib; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: celecoxib
Drug: epirubicin hydrochloride

SUMMARY:
RATIONALE: Celecoxib may stop the growth of tumor cells by stopping blood flow to the tumor. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining celecoxib with epirubicin may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of epirubicin when given together with celecoxib and to see how well it works in treating patients with hepatocellular carcinoma (liver cancer).

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of epirubicin when administered with celecoxib in patients with hepatocellular carcinoma.
* Determine the response rate in patients treated with this regimen.
* Determine the 6-month and overall survival of patients treated with this regimen.
* Determine the toxicity profile of this regimen in these patients.
* Determine the effects of this regimen on serum levels of vascular endothelial growth factor and correlate these effects with response in these patients.
* Correlate the expression of cyclooxygenase-2 in tumor tissue and nonmalignant liver tissue with response in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of epirubicin.

* Phase I:Patients receive epirubicin IV over 20 minutes on day 1 and oral celecoxib twice daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-5 patients receive escalating doses of epirubicin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 3 of 5 patients experience dose-limiting toxicity.

* Phase II: Additional patients are accrued and treated as in phase I at the MTD of epirubicin.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 3-52 patients (3-15 for phase I and 12-37 for phase II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of localized or metastatic hepatocellular carcinoma (HCC) by 1 of the following:

  * Biopsy
  * Alpha-fetoprotein (AFP) measurement (greater than 400 ng/mL if hepatitis B surface antigen [HBsAg] is negative OR greater than 1,000 ng/mL if HBsAg is positive)
* Not amenable to surgical resection or liver-directed therapy
* Measurable or evaluable disease* NOTE: *Changes in AFP alone are not sufficient
* Child-Pugh score A or B

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 75,000/mm^3

Hepatic

* Bilirubin no greater than 3.0 mg/dL
* AST no greater than 5 times upper limit of normal

Renal

* Creatinine no greater than 2.0 mg/dL

Cardiovascular

* LVEF greater than 45% by MUGA or echocardiogram

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No requirement for nonsteroidal anti-inflammatory drugs (NSAIDs) except low-dose (81 mg) aspirin
* No known hypersensitivity to aspirin or other NSAIDs
* No contraindication to cyclooxygenase-2 (COX-2) inhibitor therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No prior therapy for HCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2002-10; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of epirubicin
Response rate
Survival at 6 months
Overall survival

SECONDARY OUTCOMES:
Toxicity profile
Serum vascular endothelial growth factor levels in correlation to response
Cyclooxygenase-2 expression in tumor tissue and nonmalignant liver tissue in correlation to response

CONTACTS AND LOCATIONS:
Overall Officials: Mary Mulcahy, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States